CLINICAL TRIAL: NCT03483909
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) to Improve Gesture Control in Schizophrenia: A Randomised, Placebo-controlled, Double-blind Crossover Trial
Brief Title: Transcranial Magnetic Stimulation to Improve Gesture Control
Acronym: GestTMS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-02039
Record Dates: First submitted 2018-03-25; First posted 2018-03-30 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia and Related Disorders
Keywords: gesture; rTMS; nonverbal communication; schizophrenia; psychosis
MeSH Terms: conditions — Schizophrenia; Gestures; Nonverbal Communication; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, cross-over trial of 3 rTMS protocols
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: participants, outcome assessors and raters are blinded. rTMS application is performed by an unblinded investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- left IFG iTBS (Experimental): intermittent theta burst stimulation over the left inferior frontal gyrus
  Interventions: Device: left IFG iTBS
- right IPL cTBS (Active Comparator): continuous theta burst stimulation over the right inferior parietal cortex
  Interventions: Device: right IPL cTBS
- placebo (Placebo Comparator): Placebo TMS stimulation over the left inferior parietal cortex
  Interventions: Device: Placebo

INTERVENTIONS:
Device: left IFG iTBS — 15 daily sessions of intermittent theta burst stimulation at 80% resting motor threshold, total duration of 190 s, localization using EEG 10/20 system at F3/F4
  Arms: left IFG iTBS
Device: right IPL cTBS — 15 daily sessions of continuous theta burst stimulation at 100% resting motor threshold, total duration of 45 s, localization using EEG 10/20 system at F3/F4
  Arms: right IPL cTBS
Device: Placebo — rTMS with a placebo coil that looks identical and makes identical noises for 180 s, localization over left IPL
  Arms: placebo

SUMMARY:
The majority of schizophrenia patients is impaired in hand gesture performance, which contributes to poor functional outcome and poor communication skills. The left inferior frontal gyrus (IFG) and the left inferior parietal lobe (IPL) are key nodes of the gesture network, which is less active in patients with schizophrenia. Here, the investigators test single sessions of rTMS/TBS known to either enhance or inhibit local brain activity for app. 1 hour. The investigators aim to determine, which protocol may improve gesture performance in patients and healthy controls. This is a randomized, double-blind, cross-over, placebo-controlled single-center trial in 20 patients with schizophrenia spectrum disorders and 20 healthy controls. Gesture performance will be tested immediately after each TMS session, which are separated by 48 hours. Results of this study will inform larger interventional trials comparing 2 TMS protocols with repeated administration.

DETAILED DESCRIPTION:
Schizophrenia is associated with poor social functioning, which is perturbed by deficits in social interaction including nonverbal communication. The use of hand gestures is critical for nonverbal communication, but the majority of schizophrenia patients has severe gesture impairments. Today no intervention may ameliorate gesture impairments. Patients with gesture impairments have altered structure and function of the gesture network, particularly the left inferior frontal gyrus (IFG) and also the left inferior parietal lobe (IPL). Noninvasive brain stimulation techniques may alter local brain function. Repetitive transcranial magnetic stimulation (rTMS) and particularly theta burst stimulation (TBS) for a few mins is a very safe method to alter brain states locally for approximately 1 hour. Indeed, facilitatory stimulation of the left frontal cortex by transcranial direct current stimulation (tDCS) demonstrated improved gesture perception and interpretation in healthy subjects. In addition, inhibitory stimulation with continuous theta burst stimulation (cTBS) over left IFG may perturb gesture performance in healthy subjects. Thus, the investigators hypothesize that local changes of brain activity within the gesture network would change gesture performance. Particularly, facilitatory intermittent theta burst stimulation (iTBS) of the left IFG would improve gesture performance. The investigators will test single sessions of rTMS in healthy subjects and schizophrenia patients. If one of the protocols proves to have superior effects, this result will help to plan interventional trials targeting social interaction deficits in schizophrenia. The aim of the study is to determine the effect of one session of iTBS over the left IFG on gesture performance compared to cTBS over the right IPL (active comparator) and one placebo rTMS sessions. This is a randomized, double-blind, cross-over, placebo-controlled single-center trial in 20 patients with schizophrenia spectrum disorders and 20 healthy controls. After baseline assessment of gesture performance, participants will receive one rTMS protocol at each time point, immediately followed by assessments of gesture performance and dexterity. rTMS sessions will be separated by 48 hours. Gesture performance will be measured with video recorded Test of Upper Limb Apraxia, which is rated blindly according to a manual.

ELIGIBILITY:
Inclusion Criteria:

* Right handed according to the Edinburgh Handedness Inventory
* Ability and willingness to participate in the study
* Ability to provide written informed consent
* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Spent majority of childhood/adolescence in Switzerland
* Patients: schizophrenia spectrum disorder according to Diagnostic and Statistical Manual version 5 (DSM-5)

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Metal objects on or in the body (e.g. grenade splinter, cardiac pacemaker, vessel clips, metal prostheses, contraceptive coil, cochlear implants, hearing aid, tooth implant)
* History of neurosurgery, any severe head wounds, history of neurologic disorders impacting gesture, e.g. Parkinson's disease, stroke, multiple sclerosis sclerosis and epilepsy, convulsion or seizure
* History of any hearing problems or ringing in the ears.
* Active drug addiction except nicotine
* Controls: first-degree relatives with schizophrenia spectrum disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
Test of Upper Limb Apraxia | 10 mins after baseline assessment
  Standardized gesture performance test, video recorded and rated according to manual by a rater blind to treatment and group
Test of Upper Limb Apraxia | 10 mins after left IFG iTBS
  Standardized gesture performance test, video recorded and rated according to manual by a rater blind to treatment
Test of Upper Limb Apraxia | 10 mins after right IPL cTBS
  Standardized gesture performance test, video recorded and rated according to manual by a rater blind to treatment
Test of Upper Limb Apraxia | 10 min after placebo stimulation
  Standardized gesture performance test, video recorded and rated according to manual by a rater blind to treatment

SECONDARY OUTCOMES:
Coin rotation | 20 min after baseline assessment
  Test of dexterity, 3 trials of 10s to rotate a .5 Swiss Francs (SFr) coin between thumb, index and middle finger, video recorded, rated blindly according to number of coin half turns
Coin rotation | 20 min after left IFG iTBS
  Test of dexterity, 3 trials of 10s to rotate a .5 SFr coin between thumb, index and middle finger, video recorded, rated blindly according to number of coin half turns
Coin rotation | 20 min after right IPL cTBS
  Test of dexterity, 3 trials of 10s to rotate a .5 SFr coin between thumb, index and middle finger, video recorded, rated blindly according to number of coin half turns
Coin rotation | 20 min after placebo stimulation
  Test of dexterity, 3 trials of 10s to rotate a .5 SFr coin between thumb, index and middle finger, video recorded, rated blindly according to number of coin half turns

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Walther, MD, Principal Investigator — University of Bern, University Hospital of Psychiatry
Locations (1):
- University Hospital of Psychiatry, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share the data, because they cannot anonymize the video data sufficiently